CLINICAL TRIAL: NCT00913783
Title: Comparative, Randomized, 2-way Crossover Bioavailability Study of Geneva and Basel (Anafranil) 25 mg Clomipramine Hydrochloride Capsules In Health Adult Males Under Fasted Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Geneva and Basel (Anafranil) 25 mg Clomipramine Hydrochloride Capsules Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 920256
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Depression
Keywords: Antidepressant
MeSH Terms: conditions — Depression | interventions — Clomipramine

ARMS (2):
- 1 (Experimental): Clomipramine Hydrochloride 25 mg Capsules (Geneva Pharmaceuticals)
  Interventions: Drug: Clomipramine Hydrochloride 25 mg Capsules (Geneva Pharmaceuticals)
- 2 (Active Comparator): Anafranil Clomipramine Hydrochloride 25 mg Capsules (Basel)
  Interventions: Drug: Anafranil Clomipramine Hydrochloride 25 mg Capsules (Basel)

INTERVENTIONS:
Drug: Clomipramine Hydrochloride 25 mg Capsules (Geneva Pharmaceuticals)
  Arms: 1
Drug: Anafranil Clomipramine Hydrochloride 25 mg Capsules (Basel)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of Geneva and Basel (Anafranil) 25 mg Clomipramine Hydrochloride capsules under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 1992-11; Primary Completion 1992-12 (Actual); Study Completion 1992-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lalonde, Pharm.D., Principal Investigator — Phoenix International Life Science Inc.